CLINICAL TRIAL: NCT06810726
Title: EVALUATION OF THE SAFETY AND THE CLINICAL PERFORMANCE IN TREATMENT OF CHRONIC DIABETIC FOOT ULCER, WITH THE TROPOCELLS®, BASED AUTOLOGOUS PLATELET RICH FIBRIN (Tropocells(R) Autologous PRF Systems)
Brief Title: Evaluate Use of Tropocells(R) Autologous Platelet-rich Fibrin (PRF) for Wagner Grade 1 and Grade 2, Mild to Mod Neuroischemic Plantar Diabetic Foot Ulcer Wound Care.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Estar Medical dba Medical Technologies, LTD (Industry)
Collaborators: WCG IRB (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RND054-Tropocells PRF for DFU
Record Dates: First submitted 2025-01-17; First posted 2025-02-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot Ulcer; Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus (T2DM); Neuroischemic Foot Ulcer; Chronic Wound of the Lower Limb (Leg Ulcer or Foot Ulcer); Chronic Wound Care
Keywords: PRF used for Wagner Grade 2 DFU; Tropocells Platelet-rich Fibrin; Platelet-rich Plasma (PRP); Platelet-derived Factors for wound care; Chronic Wound Care
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Leg Ulcer; Foot Ulcer

STUDY DESIGN:
Intervention Model Description: TROPOCELLS(R) Autologous Platelet-Rich Plasma (PRF) Prospective, open-label, non-randomized, single-arm, single-agent Tropocells(R) Platelet-rich fibrin (PRF) device used to render PRF therapy applied weekly, with the primary endpoint complete (100%) wound closure response to a 12-week treatment period, where closed wounds will undergo an adjudicated assessment.
Masking Description: Validation Process- upon completion of treatment the cases will be evaluated by 3rd party validator who will review the photographs to determine if complete wound closure has occurred.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- T1DM,T2DM participants with non-infected, neuroischemic, chronic foot ulcers (Experimental): During Screen-the participant will be treated with standard of care (SOC) for 2 weeks, including education, nutritional supplement, weekly wound assessments and care with off-loading. After the two weekly visits, subjects who meet the inclusion/exclusion criterion, show adequate perfusion and area reduction less than 20%, and comply with the standard of care will be enrolled in the Active Treatment Phase. During the Active Treatment Phase, subjects will be treated weekly with TropoCells® Autologous Platelet-rich Fibrin (PRF) for twelve (12) weeks and continued SOC. Wound area will be documented with measures and photographs before and after cleansing and debridement (as needed). Clean wounds treated topically with active therapy will be covered with a non-adherent layered absorbent foam dressing with an external protective third layer. Mild compression will be applied with continued off-loading at least 2 week after closure. Follow-up evaluation after closure at 1 and 3 months.
  Interventions: Device: Platelet Rich Plasma

INTERVENTIONS:
Device: Platelet Rich Plasma — Tropocells(R) Autologous Platelet-Rich Fibrin

SUMMARY:
The goal of this investigational study is to evaluate the safety and clinical performance of Tropocells Autologous Platelet-rich Fibrin (PRF) for wound care for both males and females, ages 18-80 years old, with Grade 1 and 2, mild to moderate, neuroischemic diabetic chronic foot ulcers in subjects with Type 1 and Type 2 Diabetes Mellitus. The main question[s] it aims to answer [is/are]:

Measure 1: Wound Closure with Tropocells Autologous PRF System for DFU Measure 2: Safety of Tropocells Autologous PRF System for DFU Researchers will enroll to acquire approximately 30 evaluable subjects with no comparison group.

Run-In Phase (2 weeks): participants with chronic diabetic foot wounds will undergo a 2-week run in phase presenting to the clinic for weekly visits, for standard of care.

Active Treatment Phase (12 weeks): participants that do not show a reduction of at least 20% may be qualified to advance to the active treatment phase where wounds will be evaluated and treated weekly in the research clinic to receive standard of care with Tropocells Autologous PRF System.

Follow-up Phase (1 month and 3 months): participants with wounds that losed during the Active Treatment Phase ( 100% wound closure with two weekly assessments demonstrating persistent closure) will be advanced to the follow-up phase to show if the wound remains closed at 1 month and 3 months.

DETAILED DESCRIPTION:
Run-In Phase (2 weeks): participants with chronic diabetic foot wounds will undergo a 2-week run in phase presenting to the clinic for weekly visits, where they will receive standard of care Including-

* nutritional supplementation for 2 weeks,
* wound assessment with photos and measurements,
* wound care including cleansing and debridement,
* wound dressings,
* mild compression of the lower extremity, and
* off-loading with a removable boot.

Active Treatment Phase (12 weeks): participants that do not show a reduction of at least 20% may be qualified to advance to the active treatment phase where wounds will be evaluated and treated weekly in the research clinic. In addition to standard of care, Tropocells Autologous PRF Systems gel clot will be placed on the wound bed after cleansing and debridement prior to wound dressing and off-loading.

Data will be captured for:

Primary Outcome- Clinical Performance with complete wound closure, and Secondary Outcome(s)-

* Safety assessing adverse events (AE) and severe adverse events (SAE),
* Measures of Clinical Performance including,

  * trajectory of wound area reduction
  * percent (%) of area reduction,
  * proportion of wound area reduction

Follow-up Phase (1 month and 3 months): participants that have 100% wound closure with two weekly assessments demonstrating persistent closure, will be advanced to the follow-up phase, where they will be assessed at 1 month and 3 months with photos and measurements to show if they remain closed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Type 1 or Type 2 Diabetes
3. Grade 2, DFU, non-infected, below the ankle,1.0-12.0 cm2, present ≥ 30 day
4. Ulcer Size 1.0 cm2 to 12.0 cm2
5. Wound location will be distal to the malleolus, excluding between the toes, with no exposed capsule, tendon, or bone, and no tunneling, undermining, or sinus tracts, a depth of ≤ 5mm
6. If more than one non-healing wound is present, the selected ulcer will be the largest and ≥ 1 cm2 in size.
7. At least 2.0 cm between the index wound and other wounds.
8. Study ulcer has been present for at least 30 days and has undergone the 14-day
9. Adequate vascular perfusion of the affected limb, as defined by at least one of the following: Ankle-Brachial Index (ABI) ≥ 0.65 and ≤ 1.2, Toe Pressure (TP) ≥ 30 mmHg, Transcutaneous partial pressure of oxygen (TcPO2) ≥ 30 mmHg, or skin perfusion pressure (SPP) ≥ 30 mmHg.
10. WIFI SCORE- wound grade 1, ischemia grade 0-1, and infection grade 0)
11. Screening Period of the standard of care with 20% or less wound closure.
12. No Clinical Signs of Infection at the wound site or the affected limb.
13. Post-debridement without signs of necrotic tissue.
14. Normal Platelet count ≥ 105,000 and <450, 000 (according to CBC)
15. Hemoglobin (Hgb) ≥10 g/dL and Hematocrit (HCT) ≥ 27% (according to CBC)
16. Controlled glucose level HbA1C ≤ 12%, with active treatment being conducted to reduce the value to by a primary provider or endocrinologist
17. No Chronic Renal Failure (CRF); Estimated glomerular filtration rate (eGFR) ≥ 15
18. PT/PTT - INR between 2.0-3.0 (with blood thinners).
19. Nutritional Status with no severe protein deficiency, Pre-albumen >15 mg/dL
20. Demonstrated adequate offloading using DH Walker boot with Plastazote Insole (OR equivalent off-loading device).
21. If a female of childbearing potential, must have a negative serum or urine pregnancy test at screening and use contraception or abstinence during trial.
22. Male subjects agree to use contraception or abstinence during the trial.
23. The subject has provided written informed consent before any screening procedures and agrees to comply with study procedures and requirements.

Exclusion Criteria:

1. Life expectancy is less than 12 months.
2. Anemia Hgb ≤ 10 g/dL and HCT ≤ 27%.
3. Ulcers of other than diabetic foot pathophysiology.
4. Participation in another clinical trial involving a device or a systematically administered investigational study drug or treatment within 30 days.
5. Documented sepsis, proven with blood cultures, within 2 weeks of the trial or during the Screening Phase.
6. Soft tissue infection at the designated ulcer or the same extremity within 2 weeks of the time of screening.
7. Osteomyelitis at the designated wound site; using ESR ≥ and /or CRP ≥ 7.9 mg/d as a screen.
8. CKD Level G5: Chronic Renal Failure (CRF) sufficient to require dialysis.
9. Religious constraints to using blood products, including autologous blood.
10. Alcohol or substance abuse (other than tobacco) within 2 months before enrollment.
11. Blood-borne or communicable diseases that would likely prevent full participation in the trial (e.g., HIV, AIDs, COVID, TB).
12. Participation in another clinical trial involving a device or a systematically administered investigational study drug or treatment within 30 days of initiating the trial.
13. The subject has severe lymphedema (Stage 3) where the individual cannot lift the extremity on their own secondary to the amount of edema and fluid weight.
14. The subject is undergoing hemodialysis.
15. Subjects who are cognitively impaired, unable to understand the informed consent, or have a health care proxy.
16. Subjects with sickle cell anemia, thrombocytopenia, leukemia, or blood dyscrasia.
17. History of problems with coagulation, abnormal thrombocytes (platelets), or receiving heparin intravenously; subjects taking coumadin, aspirin, clopidogrel, or other oral anti-coagulants are not excluded.
18. Anemia where weekly blood draws of 12 or 23 per week may not be tolerated.
19. Received electrostimulation, hyperbaric treatments, growth factors, or any cell or tissue-derived therapy for any wounds 30 days before entry into the study.
20. Systemic corticosteroids, (except for subjects receiving inhaled corticosteroid treatments for asthma or COPD) 30 days before entry into the study.
21. Received within 30 days before the study or scheduled to receive medications or treatments known to interfere with or affect the rate or quality of wound closure (e.g., systemic steroids, immunosuppressive therapy, autoimmune disease therapy within the past 12 months, dialysis, radiation therapy to the treatment area, vascular surgery, angioplasty, or thrombolysis.
22. Received radiation therapy or chemotherapy within the previous 3 months.
23. Subjects with known sensitivity to blood components such as those in the PRF kit.
24. The subject has inadequate venous access for repeated blood draws required for the PRP preparation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Complete wound closure | 12 weeks of active therapy weekly applications
  * An independent validation will be performed by an independent wound care specialist who will determine if the wound is fully closed, demonstrating 100% re-epithelialization persisting for two (2) subsequent weekly assessments. The validation will be reviewed with the treating researcher and the PI to formalize the results reported to the biostatistician for analysis. The biostatistician will perform and report the following analysis.
  * Number of subjects achieving complete epithelialization at 12 weeks in the Intent to Treat (ITT) population.
  * Number of subjects achieving complete epithelialization at 12 weeks in the Per Protocol (PP) population.

SECONDARY OUTCOMES:
Safety- Adverse Events, Serious Adverse Events, Deviations, Violations | Screening Phase- 2 weeks and Active Treatment Phase- 12 weeks
  The biostatistician will measure and report:
  1. Adverse Events (AE), including any untoward or unfavorable medical occurrence in a human study participant, including any abnormal sign (e.g. abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with a participant's involvement in the research, whether or not considered related to participation in the research, and
  2. Serious Adverse Events (SAE), including any adverse event that: i) results in death, ii) is life-threatening, or places the participant at immediate risk of death from the event as it occurred, iii) requires or prolongs hospitalization, iv) causes persistent or significant disability or incapacity,and/o v) results in congenital anomalies or birth defects vi) Is another condition which in the investigator's judge to represent significant hazards, and 3) Unanticipated Problem (UP):
  Defined by DHHS 45 CFR part 46 as any incident, experience, or outcome that meets the criteria.

OTHER OUTCOMES:
Percentage Area Reduction (PAR) | 12 weeks
  percent wound closure compared to baseline (beginning Active Treatment Phase) to complete wound closure performing assessments every two weeks during the Active Treatment Phase (weeks: 2, 4, 6, 8, 10, and 12).
Time to Wound Closure | 12 weeks
  Active Phase week (0) will be compared to the week of closure. All weeks will be followed for 2 weekly visits after closure. Closure noted at the last Active Phase visit will be followed for 2 additional weeks to ensure proper documentation of closure.

CONTACTS AND LOCATIONS:
Overall Officials: Adrianne P Smith, MD, Study Director — Sanogenix Medical, LLC; Marcus L. Gitterle, MD, Principal Investigator — WoundCentrics
Locations (2):
- United States (2):
  - WoundCentrics Wound Care & Hyperbarics -Corpus Christi - Shoreline, Corpus Christi, Texas
  - Woundcentrics Wound Care Center At Corpus Christi South, Corpus Christi, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) will be shared with the organizations used to analyze the data (Strategic Solutions, Inc) and to present the data to the FDA/CBER for the 510K Submission.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anticipated 510K submission- Jul2026 Duration while 510K is under consideration- 90 days
Access Criteria: The clinical research organization, Global Clinical Research Institute-GCRI), and biostatistician (Strategic Solutions, Inc.), regulatory consultant, Biologics Consulting Group-BCG,and the WCG IRB will be able to access the data in deidentified format and potentially as individual patient data (IPD) during trial conduct or in preparation for the 510K submission.
  If the FDA clears the device, we may publish the results to share with the medical community; however, only deidentified case studies and/or analyzed data will be used.
  IPD may also be shared with other researchers in a registry once the device has been cleared.
URL: https://www.wcgclinical.com/wp-content/uploads/2020/08/Guide_for_Researchers-1.pdf?v=1709839112

REFERENCES:
- [Background] Piccin A, Di Pierro AM, Canzian L, Primerano M, Corvetta D, Negri G, Mazzoleni G, Gastl G, Steurer M, Gentilini I, Eisendle K, Fontanella F. Platelet gel: a new therapeutic tool with great potential. Blood Transfus. 2017 Jul;15(4):333-340. doi: 10.2450/2016.0038-16. Epub 2016 Jul 25. PMID 27483482
- [Background] Chen P, Vilorio NC, Dhatariya K, Jeffcoate W, Lobmann R, McIntosh C, Piaggesi A, Steinberg J, Vas P, Viswanathan V, Wu S, Game F. Guidelines on interventions to enhance healing of foot ulcers in people with diabetes (IWGDF 2023 update). Diabetes Metab Res Rev. 2024 Mar;40(3):e3644. doi: 10.1002/dmrr.3644. Epub 2023 May 25. PMID 37232034